CLINICAL TRIAL: NCT05542524
Title: Oral Care of Patients Treated With Anti-RANK-ligand Antibodies for a Giant Cell Tumour: Retrospective Study at the University Hospitals of Strasbourg
Brief Title: Oral Care of Patients Treated With Anti-RANK-ligand Antibodies for a Giant Cell Tumour
Acronym: DENO
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8699
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Giant Cell Tumors
Keywords: Giant Cell Tumors; Anti-RANK-ligand antibodies
MeSH Terms: conditions — Giant Cell Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Giant cell tumors are mostly benign tomoral processes, most often responsible for areas of osteolysis in the metaphysoepiphyseal area of long bones, representing 5-6% of primary bone tumors. The bone weakening induced by these beaches leads to pain and risk of fracture, and this is what leads the patient to consult.

These tumors are found particularly in the young adult population between 20 and 40 years old, are locally aggressive, but malignant transformations and metastases (pulmonary) are quite rare.

In this study, the investigators wish to retrospectively study the oral care of patients who presented with a giant cell tumor and were treated with Denosumab at the University Hospital of Strasbourg and their associated oral follow-up

ELIGIBILITY:
Inclusion criteria:

* Adult subject, having presented a giant cell tumor treated with adjuvant or neoadjuvant denosumab at the HUS from 01/01/2014 to 08/31/2022.
* Subjects who have not expressed their opposition to the reuse of their data for scientific research purposes.

Exclusion criteria:

* Subject having expressed their opposition to the retrospective reuse of their data for scientific research purposes
* Pathology finally labeled other than giant cell tumour.
* Treatment with denosumab was not initiated because of death, change in treatment protocol, etc.
* Absence of oral follow-up element.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subject, having presented a giant cell tumor treated with adjuvant or neoadjuvant denosumab at the HUS from 01/01/2014 to 08/31/2022.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Number of Decayed, Missing, and Filled Permanent Teeth (DMFT) | Files analysed retrospectively from from January 01, 2014 to August 31, 2022 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine et Chirurgie Bucco-Dentaires - CHU de Strasbourg - France, Strasbourg, France